CLINICAL TRIAL: NCT03706222
Title: The Real World Analysis of Drug-Drug Interactions of Grazoprevir/Elbasvir in Treatment of Chronic Hepatitis C Patients in Taiwan
Brief Title: Drug-Drug Interactions of Grazoprevir/Elbasvir in Taiwan
Status: Completed | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Pin-Nan Cheng, Associate Professor, National Cheng-Kung University Hospital
Other Study IDs: MISP#57751
Record Dates: First submitted 2018-10-08; First posted 2018-10-15 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Drug Interaction Potentiation
MeSH Terms: interventions — elbasvir-grazoprevir drug combination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Drug interaction of Elbasvir/Grazoprevir: Patients treated with elbasvir/grazoprevir will be enrolled. DDI will be evaluated.
  Interventions: Drug: elbasvir/grazoprevir

INTERVENTIONS:
Drug: elbasvir/grazoprevir — Comedications during elbasvir/grazoprevir will be recorded and analyzed for potential drug-drug interaction.
  Other Names: Zepatier

SUMMARY:
Co-morbid diseases often present in a substantial proportion of patients with chronic hepatitis C (CHC) and require drugs to treat and control. Grazoprevir/elbavir is metabolized by cytochrome P-450 enzyme of liver. Drug-drug interactions (DDIs) are important issue before commencing direct acting antiviral agents (DAA) treatment for CHC patients. Few studies from Western countries reported that the percentages of DDIs of grazoprevir/elbasvir are limited.In Asia, real-world analysis of DDIs of grazoprevir/elbasvir is lacking and needs to be clarified.

DETAILED DESCRIPTION:
This is a multi-center, retrospective study. Five hospitals in Taiwan and 400 patients Patients treated with grazoprevir/elbasvir during August 2017 to July 2018 are candidates of study subjects. All the required study information will be recorded with detailed chart review.

DDI will be evaluated by HEP Drug Interactions (www.hep-druginteractions.org) assessment of comidications: Category 0: Classification not possible due to lack of information; Category 1: No clinical interaction possible; Category 2: May require dose adjustment/closer monitoring; Category 3: Coadministration not recommended or contraindicated.

The assessment of DDI will be evaluated and recorded according to the suggested categories, the number of patients at risk for a clinically relevant DDI, and the ratio of patients with at least one predicted DDI between medication of grazoprevir/elbasvir will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with grazoprevir/elbasvir are candidates of study subjects.

Exclusion Criteria:

* none

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients infected with genotype 1 or 4 hepatitis C virus and treated with elbasvir/grazoprevir during August 2017 to July 2018 in Taiwan.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2019-02-25 (Actual)

PRIMARY OUTCOMES:
the potential drug drug interaction of elbasvir/grazoprevor | DDI will be assessed before and through the 12 weeks or 16 weeks of elbasvir/grazoprevir treatment
  the ratio of patients with at least one predicted DDI will be analyzed.

SECONDARY OUTCOMES:
the comorbid diseases of CHC patients in Taiwan | Comorbid diseases will be assessed before elbasvir/grazoprevir treatment.
  Comorbid diseases will be recorded and categorized by involved organ systems before elbasvir/grazoprevir treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Pin-Nan Cheng, M.D., Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu CJ, Tseng KC, Lo CC, Tseng IH, Cheng PN. Limited drug-drug interaction of elbasvir/grazoprevir for chronic hepatitis C. J Formos Med Assoc. 2020 May;119(5):933-940. doi: 10.1016/j.jfma.2019.09.011. Epub 2019 Oct 5. PMID 31594667

DOCUMENTS (1):
  • Study Protocol (2018-07-28): https://cdn.clinicaltrials.gov/large-docs/22/NCT03706222/Prot_000.pdf